CLINICAL TRIAL: NCT00809523
Title: A Multicenter, Randomized Controlled Trial of Negative Ion Generation Versus Light-Emitting Diode Phototherapy for Seasonal Affective Disorder (SAD)
Brief Title: A Trial of Negative Ion Generation Versus Light-Emitting Diode Phototherapy for Seasonal Affective Disorder (SAD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The Litebook Company Ltd. (Industry); University of British Columbia (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Harvard University (Other); University of Toronto (Other); Clinical Associates Research, Maryland (Network); Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0810004322
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-01

CONDITIONS: Seasonal Affective Disorder
Keywords: SAD; winter depression
MeSH Terms: conditions — Seasonal Affective Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inactivated negative ion generator (Experimental): Equivalent exposure to inactivated Negative Ion Generator
  Interventions: Device: Negative Ion Generator
- LED light treatment device (Experimental): Light-emitting photodiode light treatment device, used for 30 min before 8 am
  Interventions: Device: Light-emitting Photodiode light treatment device

INTERVENTIONS:
Device: Negative Ion Generator — Equivalent exposure to inactivated Negative Ion Generator
  Arms: Inactivated negative ion generator
Device: Light-emitting Photodiode light treatment device — Light-emitting Photodiode light treatment device, used for 30 min before 8 am
  Arms: LED light treatment device

SUMMARY:
This is a randomized, controlled clinical trial of inactivated negative ion generation or light-emitting photodiode therapy for Seasonal Affective Disorder (SAD, winter depression), for subjects with a DSM IV diagnosis of Major Depression, with Seasonal Pattern, Winter type, to examine efficacy of treatments for this condition. The trial has a 1 week baseline phase and a 4 week treatment phase.

DETAILED DESCRIPTION:
This is a randomized, controlled clinical trial comparing an inactivated negative ion generation (placebo condition) and light-emitting photodiode therapy (active condition), for Seasonal Affective Disorder (SAD, winter depression), for subjects with a DSM IV diagnosis of Major Depression, with Seasonal Pattern, Winter type, to examine efficacy of treatments for this condition. Exclusion criteria included any other current treatment for SAD, as well as bipolar disorder, type 1, a chronic psychotic disorder, or a substance use not if full remission for at least one year. The trial has a 1 week baseline phase and subjects were seen weekly during a 4 week treatment phase. The study was double-blind. The study was conducted at 8 sites in the US, Canada and The Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Seasonal Affective Disorder
* Age 18 to 65

Exclusion Criteria:

* Psychotropic medication treatment
* History of light treatment for SAD
* History of mania or psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Desan, MD, PhD, Principal Investigator — Yale University; Raymond Lam, MD, Principal Investigator — University of British Columbia, Vancouver, Canada
Locations (8):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - Capital Clinical Research Associates, Rockville, Maryland
  - McLean Hospital/Harvard, Belmont, Massachusetts
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - St. John Regional Hospital, Saint John, New Brunswick
  - CAMH/University of Toronto, Toronto, Ontario
  - Sleep and Alertness Inc, Toronto, Ontario
- University Medical Center Groningen, Groningen, RB, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- LED Phototherapy Device: Light-emitting photodiode light treatment device, used for 30 min before 8 am
Period: Overall Study
Arm/Group | Inactivated Negative Ion Generator | LED Phototherapy Device
Started | 54 | 52
Completed | 47 | 48
Not Completed | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inactivated Negative Ion Generator | LED Phototherapy Device | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 52 | 106
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 38 | 80
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38
  Netherlands | 8 | 9 | 17
  Canada | 26 | 25 | 51

OUTCOME MEASURES:

1. Secondary Outcome: SIGH SAD Depression Rating
Description: SIGH SAD Structured Interview Guide for the Hamilton Depression Rating Scale, Seasonal Affective Disorder (SAD)version. This is a structured interview, which is an interview in which the clinician is provided exact questions to use to inquire about symptoms of depression and explicit standards for rating the intensity of each symptom item. The interview assesses the symptoms which make up the Hamilton Depression Rating Scale, which is the standard in the majority of clinical trials in depression. The items are augmented with additional items to reflect better the atypical depressive symptoms usually seen in SAD, eg, increased sleep, weight, appetite and fatigue. On this scale, higher scores reflect increased depression intensity. The maximum score attainable is 63, and the minimum is 0. A score of less than 9 is regarded as consistent with normal mood, the absence of major depression.
Time Frame: Weekly
Population: Intent to treat analysis last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inactivated Negative Ion Generator | LED Phototherapy Device
Number analyzed (Participants) | 54 | 52
units on a scale
  Randomization | 28.6 (6.7) | 27.7 (4.8)
  Week 1 | 23.6 (8.7) | 20.9 (7.0)
  Week 2 | 19.9 (9.3) | 17.4 (7.8)
  Week 3 | 18.6 (9.7) | 15.8 (8.3)
  Week 4 | 17.9 (10.2) | 13.3 (9.2)

2. Secondary Outcome: Clinical Global Impression of Severity
Description: The Clinical Global Impression of Severity is a 7-point scale in which the clinician gives an overall impression of depression severity, with the following anchor points: (1)Normal, not at all ill, (2)Borderline ill, (3) Mildly ill, (4)Moderately ill, (5) Markedly ill, (6)Severely ill, and (7)Among the most severely ill patients. The minimum is therefore 1 and the maximum is 7, which represents very severe depression.
Time Frame: Randomization and at 4 weeks
Population: intent to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inactivated Negative Ion Generator | LED Phototherapy Device
Number analyzed (Participants) | 54 | 52
units on a scale
  Randomization | 4.2 (0.6) | 4.2 (0.7)
  Week 4 | 3.0 (1.3) | 2.4 (1.2)
Statistical Analysis 1: Comparison: Inactivated Negative Ion Generator vs LED Phototherapy Device; Data were analyzed at the follow up timepoint (4 weeks) to test for differences between the experimental groups; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

3. Primary Outcome: Percentage Change SIGH SAD Depression Rating
Description: SIGH SAD Structured Interview Guide for the Hamilton Depression Rating Scale, Seasonal Affective Disorder (SAD)version. The items are augmented with additional items to reflect better the atypical depressive symptoms usually seen in SAD, eg, increased sleep, weight, appetite and fatigue. On this scale, higher scores reflect increased depression intensity. The maximum score attainable is 63, and the minimum is 0. A score of less than 9 is regarded as consistent with normal mood, the absence of major depression.
  Calculated: SIGH SAD score at trial end - SIGH SAD score at randomization x 100 / SIGH SAD score at randomization
Time Frame: 4 weeks
Population: Intent to treat analysis last observation carried forward.
Measure: Mean (Standard Deviation); unit: percentage of change on SIGH SAD
Arm/Group | Inactivated Negative Ion Generator | LED Phototherapy Device
Number analyzed (Participants) | 54 | 52
percentage of change on SIGH SAD | -36.4 (34.9) | -52.7 (31.7)
Statistical Analysis 1: Comparison: Inactivated Negative Ion Generator vs LED Phototherapy Device; Test type: Superiority or Other; p = 0.014, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Inactivated Negative Ion Generator | LED Phototherapy Device
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 1/54 | 7/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inactivated Negative Ion Generator (N=54) | LED Phototherapy Device (N=52)
Eye strain/glare (Nervous system disorders) | 0 (0) | 3 (3)
headache (Nervous system disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No